CLINICAL TRIAL: NCT02170402
Title: Study to Evaluate Efficacy and Safety of ADVATE in the Treatment of Previously Treated Patients With Hemophilia A
Brief Title: China ADVATE PTP Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 061301
Record Dates: First submitted 2014-06-20; First posted 2014-06-23 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human; Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Previously Treated Patients (PTPs) (Experimental): PTPs will participate sequentially with:
  Part 1: Pharmacokinetic parameters of ADVATE measured in subset of 24 participants, consisting of:
  * 12 adults (>12 years of age)
  * 12 children (≤12 years of age)
  Part 2: On-demand treatment with ADVATE for 6 months
  Part 3: Prophylaxis regimen with ADVATE for 6 months
  Interventions: Biological: Octocog alfa (recombinant human coagulation factor VIII)

INTERVENTIONS:
Biological: Octocog alfa (recombinant human coagulation factor VIII) — * Part 1: Pharmacokinetic (PK) analysis - Subset of 24 participants
  * Part 2: On-demand treatment regimen
  * Part 3: Prophylaxis treatment regimen
  Other Names: ADVATE

SUMMARY:
The purpose of this study is to assess efficacy, safety and pharmacokinetics of ADVATE in the treatment and prevention of bleeding episodes (BEs)

ELIGIBILITY:
Main Inclusion Criteria:

* Ethnic Chinese
* is of any age
* has a documented diagnosis of severe or moderately severe hemophilia A (congenital FVIII deficiency: baseline Factor VIII (FVIII) ≤ 2%)
* has documented and verified >50 exposure days (EDs) to FVIII (recombinant or plasma derived)
* is receiving on-demand treatment with FVIII at the time of enrolment in this study
* has negative history of inhibitor development
* is HIV negative or HIV positive with stable disease and CD4+ count ≥ 200 cells per mm^3
* is negative for Hepatitis C virus (HCV); Or participant is HCV positive with chronic stable hepatitis as assessed by investigator

Main Exclusion Criteria:

* has prior history of hypersensitivity or anaphylaxis associated with receipt of FVIII
* is diagnosed with other bleeding disorder(s) other than hemophilia A, including but not limited to thrombocytopenia (platelet count < 100000 /mL)
* has been exposed to an investigational product (IP) within 30 days prior to the screening visit or is scheduled to participate in another clinical study involving an IP or investigational device during participation in the study
* is planned, or likely to have surgery during the study period
* has end-stage renal failure or evidence of a severe or uncontrolled systemic disease as judged by the investigator
* has active hepatic disease (alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels > 5 times the upper limit of normal)
* has clinical or laboratory evidence of severe liver impairment including (but not limited to) a recent & persistent international normalized ratio (INR) >1.4, and/or the presence of splenomegaly and/or significant spider angioma on physical exam, and/or a history of esophageal hemorrhage or documented esophageal varices
* is a family member of the investigator or site staff

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-06-26 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Percentage of reduction in annualized bleed rate (ABR) during prophylactic treatment compared to ABR during on demand treatment | 12 months
  Computed as:
  {[median ABR on-demand - median ABR prophylaxis]÷[median ABR on-demand]}*100%
  The ABR, will be assumed to have a negative binomial distribution. The 2 treatment regimens (on-demand and prophylaxis) will be compared in terms of mean ABR within a generalized linear model framework (with a logarithmic link function which is the default for the negative binomial distribution), accounting for the fixed effect of study arm and the follow-up time (in years) as an offset. Ratios between treatment means (95% CI) will be estimated within this model.

SECONDARY OUTCOMES:
Number of units per kg body weight of ADVATE required to resolve a bleeding episode (BE) | 12 months
Number of infusions of ADVATE required to resolve a bleeding episode (BE) | 12 months
Overall evaluation of efficacy on a four-point scale (Excellent-Good-Fair-Poor) | 12 months
Annualized bleeding episode rates (ABR) according to bleed type and bleed etiology summarized by treatment regimen | 12 months
  Bleed types and etiologies summarized by treatment regimen (prophylaxis, on-demand) including:
  * Joint bleeds
  * Non-joint bleeds
  * Spontaneous bleeds
  * Traumatic bleeds
  * Target joint bleeds
Inhibitor incidence | 13 months
  Inhibitor incidence in:
  1. Previously treated patients (PTPs) with previous 51-150 exposure days (EDs) to Factor VIII (FVIII)
  2. PTPs with previous >150 EDs to FVIII
Adverse events according to relatedness, seriousness, and severity | 13 months
Area under the plasma concentration/time curve from time 0 to infinity | Within 30 minutes prior to the start of the infusion through 48 hours post-infusion
  Computed as AUC0-t + Ct/ λz, where t is the time of last quantifiable concentration, Ct is the last quantifiable concentration, and λz is the terminal rate constant
Mean Residence Time (MRT) | Within 30 minutes prior to the start of the infusion through 48 hours post-infusion
  Computed as AUMC0-∞ / AUC0-∞ - TI/2, where AUMC0-∞ will be determined in a similar manner as AUC0-∞ and TI represents infusion duration [hour]
Clearance (CL) | Within 30 minutes prior to the start of the infusion through 48 hours post-infusion
  Computed as Dose/ AUC0-∞
Incremental Recovery (IR) at Cmax | Within 30 minutes prior to the start of the infusion, and within 1 hour post-infusion
  Computed as: (Cmax - Cpre-infusion)/Dose, where Cmax will be determined as the highest concentration achieved within one hour after infusion
Elimination phase half-life | Within 30 minutes prior to the start of the infusion through 48 hours post-infusion
  Computed as: ln2/ λz. λz will be estimated from the slope of natural log-linear fitting to latter quantifiable concentrations, with largest adjusted R^2
Volume of distribution at steady state (Vss) | Within 30 minutes prior to the start of the infusion through 48 hours post-infusion
  Computed as: CL * MRT

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (11):
- China (11):
  - Peking Union Medical College Hospital, Dongcheng, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Tongji Hosp, Tongji Med. Col, Huazhong Univ. of Sci. & Tech/ Wuhan Union Hospital, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College of Hongzhong Science and Techology University, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of College of Medicine, Zhengjiang University, Hangzhou, Zhejiang
  - Beijing Children's Hospital Affiliated to Capital University of Medical Sciences, Beijing
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Hospital of Blood Disease, Chinese Academy of Medical Sciences, Tianjin